CLINICAL TRIAL: NCT01776684
Title: Detection of Resistance Genes From Serially Collected Plasma DNA in Non-small Cell Lung Cancer Patients Harboring EGFR Activating Mutation Who Are Being Treated With EGFR TKIs
Brief Title: Evaluation of EGFR TKI Resistance Mechanism Using Plasma DNA Analysis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Myung-Ju Ahn, M.D., Professor, Samsung Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2011-10-054
Record Dates: First submitted 2013-01-23; First posted 2013-01-28 (Estimated); Last update posted 2013-01-28 (Estimated); Status verified 2013-01

CONDITIONS: EGFR Mutation Positive Non-small Cell Lung Cancer
MeSH Terms: interventions — Gefitinib; Erlotinib Hydrochloride; Afatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EGFR positive arm (Experimental): Patients with NSCLC harboring activating EGFR mutation (deletion in exon 19, L858R mutation in exon 21)
  Interventions: Drug: EGFR TKIs (gefitinib, erlotinib, afatinib, et al)

INTERVENTIONS:
Drug: EGFR TKIs (gefitinib, erlotinib, afatinib, et al)

SUMMARY:
To detect resistance gene from serially collected plasma DNA in non-small cell lung cancer harbouring EGFR activating mutation who are being treated with EGFR TKIs by using castPCR method.

ELIGIBILITY:
Inclusion Criteria:

* 1. Histologically confirmed NSCLC 2. Aged of or older than 20 years 3. ECOG performance status 0-2 4. Adequate hematological, renal, hepatic function 5. Patients with tumors harboring EGFR mutation (del 19 or L858R mutation) 6. Patient who are about to be treated with EGFR TKI (gefitinib, erlotinib or other EGFR TKI) 7. At least more than one measurable disease 8. Informed consent

Exclusion Criteria:

* 1. Active infection 2. Active bleeding

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2012-06; Primary Completion 2014-05 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
detection of resistant gene | 24 months
  To evaluate the efficiency of castPCR method for detection of resistance genes, especially, T790M mutation from serially collected plasma DNA in non-small cell lung cancer patients harboring EGFR activating mutation who are being treated with EGFR TKIs

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea